CLINICAL TRIAL: NCT00424034
Title: Phase I Study of Ambrisentan - Single Dose Study in Healthy Japanese Male Subjects
Brief Title: A Study of GSK1325760A in Healthy Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMB107623
Record Dates: First submitted 2007-01-16; First posted 2007-01-18 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Subjects
Keywords: safety; Pharmacokinetics; effect of food on pharmacokinetics
MeSH Terms: interventions — ambrisentan

INTERVENTIONS:
Drug: GSK1325760A

SUMMARY:
To investigate the safety, tolerability, pharmacokinetics and the effect of food on pharmacokinetics after single oral administrations of GSK1325760A

DETAILED DESCRIPTION:
Phase1 study of GSK1325760A

- A double blind, single center, randomised, placebo-controlled, partially crossover, single dose study to investigate the safety, tolerability, pharmacokinetics and to assess the effect of food on pharmacokinetics of ascending oral doses of GSK1325760A in healthy Japanese male subject -

ELIGIBILITY:
Inclusion Criteria:

* They are considered as healthy by the investigator at screening. Healthy subjects are defined as individuals who are free from clinically significant illness or disease as determined by their medical history, physical examination, clinical laboratory tests, vital sign, 12-lead ECG, immunology tests and urinary drug screening tests.
* They are Japanese males.
* Aged 20 to 64 years, inclusive.
* They have a body mass index (weight/height2) at screening in the range of 18.5 and <25.0 kg/m2 inclusive. Standard weight is in the range of 55-85 kg inclusive.
* Blood pressure and pulse rate at screening within the normal range (systolic 90-140 mmHg, diastolic 40-90 mmHg, pulse rate 40-90bpm).
* They have the following clinical laboratory test
* Biochemistry (AST(GOT), ALT(GPT), ALP, LDH and gamma-GTP : within normal range at screening.
* Haematology (RBC, Hb and Ht) below upper limit normal range at screening.
* Normal ECG at screening (QTc value of <440msec).
* They give their consent to be able to abstain from sexual intercourse or use condom for contraception from at screening until post-study screen.
* They are capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* They are non-smokers (at least 6 months).
* They are able to attend all visits and complete the study.

Exclusion Criteria:

* The subject has any clinically relevant abnormality on medical examination, vital sign, clinical laboratory test or medical history at screening in the medical opinion of the investigator or the subject has a medical history that is not considered as eligible for inclusion in this study by the investigator.
* The subject has an allergy for any drug or idiosyncrasy. This excludes a pollen allergy without current symptoms.
* The subject has participated in a clinical study or post-marketing study with an investigational or a non-investigational product or device during the previous 4 months of the first dosing.
* The subject is concurrently participating in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational product or device.
* The subject is positive for syphilis, HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody.
* The subject is positive for urine drugs of abuse test.
* The subject has donated a unit of blood (>400mL) within the previous 4 months or (>200mL) within the previous 1 month of screening.
* The subject is currently taking regular (or a course of) medication (including prescribed drug, over-the-counter medication and herbal preparations). Medication nor permitted during the study must be discontinued 14 days prior to dosing.
* The subject has a history or current conditions of drug abuse or alcoholism according to ICD10.
* The subject has a history of regular alcohol consumption exceeding 7 drinks/week (1 drink = 350mL of beer) within 6 months of the first dosing.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Adverse events Change in Clinical laboratory test Vital sign 12-lead ECG Plasma concentration Urine concentration | on 5 or 6 days after dosing

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline